CLINICAL TRIAL: NCT00110071
Title: A Clinical Trial Evaluating I131-Tositumomab (Anti-CD20) With Escalating Doses of Fludarabine Followed by Autologous or Syngeneic Stem Cell Transplantation for Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma in Patients 60 Years of Age and Older
Brief Title: Iodine I 131 Tositumomab and Fludarabine Phosphate in Treating Older Patients Who Are Undergoing an Autologous or Syngeneic Stem Cell Transplant for Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1943.00; NCI-2009-01470 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA044991 (NIH)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — fludarabine phosphate; Peripheral Blood Stem Cell Transplantation; tositumomab I-131; Flow Cytometry; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemoradioimmunotherapy) (Experimental): Patients receive a dosimetric dose of iodine I 131 tositumomab IV over 40-60 minutes on day -24 followed by gamma camera imaging over the next 6 days. Patients then receive a therapeutic dose of iodine I 131 tositumomab via central line over 40-60 minutes on day -14. Patients also receive fludarabine phosphate IV QD on days -11 to -9 OR days -11 or -7. Patients undergo autologous or syngeneic peripheral blood stem cell transplantation on day 0.
  Interventions: Drug: fludarabine phosphate; Procedure: peripheral blood stem cell transplantation; Radiation: iodine I 131 tositumomab; Other: laboratory biomarker analysis; Other: flow cytometry; Genetic: polymerase chain reaction

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Procedure: peripheral blood stem cell transplantation — Undergo transplantation (infusion of autologous or syngeneic PBSC via central line)
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Radiation: iodine I 131 tositumomab — Given IV (dosimetric dose) or via central line (therapeutic dose)
  Other Names: 131-I-anti-B1 antibody; 131-I-anti-B1 monoclonal antibody; I131-MOAB-B1; iodine I 131 MOAB anti-B1; iodine I 131 monoclonal antibody anti-B1
Other: laboratory biomarker analysis — Correlative studies
Other: flow cytometry — Correlative studies
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR

SUMMARY:
This phase I trial studies the side effects and best dose of fludarabine (fludarabine phosphate) when given together with iodine I 131 tositumomab in treating older patients who are undergoing an autologous or syngeneic stem cell transplant for relapsed or refractory B-cell non-Hodgkin's lymphoma (NHL). Radiolabeled monoclonal antibodies, such as iodine I 131 tositumomab, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. A peripheral stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy and radiation therapy. Giving iodine I 131 tositumomab together with fludarabine followed by autologous stem cell transplant may be an effective treatment for NHL

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximally tolerated dose of fludarabine that can be combined with 131I-anti-CD20 (iodine I 131 tositumomab) delivering =< 27Gy to critical normal organs followed by autologous or syngeneic transplantation in patients >= 60 years of age with relapsed B-NHL.

SECONDARY OBJECTIVES:

I. To assess the overall and progression-free survival of the above regimen in such patients.

II. To evaluate the response rates of the above therapy.

III. To evaluate the toxicity and tolerability of the above therapy.

IV. To evaluate the feasibility of delivering concurrent high-dose radioimmunotherapy (RIT) and chemotherapy.

OUTLINE: This is a dose-escalation study of fludarabine phosphate as used in combination with I 131 tositumomab and stem cell transplant.

Patients receive a dosimetric dose of iodine I 131 tositumomab intravenously (IV) over 40-60 minutes on day -24 followed by gamma camera imaging over the next 6 days. Patients then receive a therapeutic dose of iodine I 131 tositumomab via central line over 40-60 minutes on day -14. Patients also receive fludarabine phosphate IV once daily (QD) on days -11 to -9 OR days -11 or -7. Patients undergo autologous or syngeneic peripheral blood stem cell transplantation on day 0.

Patients with circulating lymphoma cells by peripheral smear receive tositumomab IV over 1 hour OR rituximab IV over 1 hour followed by tositumomab IV over 1 hour before the dosimetric iodine I 131 tositumomab infusion.

After completion of study treatment, patients are followed up at 1, 3, 6, and 12 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of lymphoma expressing the CD20 antigen and generally must have failed at least one prior standard systemic therapy; the exception will be mantle cell lymphoma (MCL) patients, who may be enrolled while in first complete remission (CR) in accordance with current transplant standard of care for these patients
* Creatinine (Cr) < 2.0
* Bilirubin < 1.5 mg/dL, with the exception of patients thought to have Gilbert's syndrome, whom may have a total bilirubin above 1.5 mg/dL
* All patients eligible for therapeutic study must have (>= 2x10^6 CD34/kg) autologous hematopoietic stem cells harvested and cryopreserved, or this number of cells harvested from a syngeneic donor
* Patients must have an expected survival of > 60 days and must be free of major infection
* DONOR: Syngeneic donors must be confirmed syngeneic by ABO typing, human leukocyte antigen (HLA) typing, and variable number tandem repeat (VNTR) analysis
* DONOR: Syngeneic donors must meet eligibility under Standard Practice Guidelines/Standard Treatment

Exclusion Criteria:

* Circulating anti-mouse antibody (HAMA) (to be determined before both dosimetry and therapy)
* Systemic anti-lymphoma therapy given in the previous 30 days before the scheduled therapy dose
* Inability to understand or give an informed consent
* Prior radiation > 20 Gy to any critical normal organ (e.g., lung, liver, spinal cord, > 25% of red marrow)
* Central nervous system lymphoma
* Other serious medical conditions considered to represent contraindications to bone marrow transplant (BMT) (e.g., abnormally decreased cardiac ejection fraction, diffusing capacity (DLCO) < 50% predicted, patient on supplemental oxygen, acquired Immunodeficiency syndrome [AIDS], etc.)
* Pregnancy
* Prior bone marrow or stem cell transplant
* South West Oncology Group (SWOG) performance status >= 2
* Unable to perform self-care during radiation isolation
* Patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma/well differentiated lymphocytic lymphoma

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-01; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose/dose limiting toxicity | Up to 30 days post-transplant
  Assessed according to Bearman scale for Regimen-Related Toxicities.

SECONDARY OUTCOMES:
Overall and progression-free survival rate | Up to 6 years
Response rate | Up to 12 months
Toxicity/tolerability of study regimen | Through day 100 post-transplant
  Type, frequency, and severity of adverse events grade 3 and above (assessed by National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) v3.0.
Feasibility of concurrent high-dose radioimmunotherapy and chemotherapy | Through day -7 prior to transplant
  Ability to administer complete course of I 131-tositumomab and fludarabine phosphate as descried in protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Gopal AK, Gooley TA, Rajendran JG, Pagel JM, Fisher DR, Maloney DG, Appelbaum FR, Cassaday RD, Shields A, Press OW. Myeloablative I-131-tositumomab with escalating doses of fludarabine and autologous hematopoietic transplantation for adults age >/= 60 years with B cell lymphoma. Biol Blood Marrow Transplant. 2014 Jun;20(6):770-5. doi: 10.1016/j.bbmt.2014.02.004. Epub 2014 Feb 12. PMID 24530971